CLINICAL TRIAL: NCT03526198
Title: Quantification of Distribution of the Mass Center for a Controlled Force Platform Reaction to the Ground
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cruzeiro do Sul (Other)
Responsible Party: Principal Investigator, Leandro Lazzareschi, PhD, University of Mogi das Cruzes
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 56483816.8.0000.5497
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Balance
Keywords: Force plate; Center of mass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (adult) (Experimental): Each volunteer stood on the platform. The duration of the tests was standardized at 10 seconds for each angulation variant of the test. The tilt variables occurred every 5 degrees oscillating in the two-dimensional movement of the ankle joint. The test was discontinued when the volunteer failed to remain balanced at the tested angulation for more than 10 seconds (thus shifting the foot (s) from the initial position or supporting with one and / or both arms at the therapist or at the support bars ) or when it reached maximum angulation
  Interventions: Device: Force plate
- Group 2 (elderly) (Experimental): Each volunteer stood on the platform. The duration of the tests was standardized at 10 seconds for each angulation variant of the test. The tilt variables occurred every 5 degrees oscillating in the two-dimensional movement of the ankle joint. The test was discontinued when the volunteer failed to remain balanced at the tested angulation for more than 10 seconds (thus shifting the foot (s) from the initial position or supporting with one and / or both arms at the therapist or at the support bars ) or when it reached maximum angulation
  Interventions: Device: Force plate

INTERVENTIONS:
Device: Force plate — Device: force plate An equipment model with the approach of providing the evaluated person with the movement that is closest to the biomechanical and functional reality of the ankle and foot joint and which could equalize the possible changes of the center of mass would contribute to the clinical evaluation and would provide a more efficient therapeutic reasoning rehabilitation.

SUMMARY:
This study developed a controlled soil reaction force platform that provided controlled mechanical stimuli to quantify the distribution of the center of mass as a function of the angular variation of the ankle in the elderly in the upright position.

DETAILED DESCRIPTION:
Usually the balance evaluation the center of mass displacement for the analysis of postural control is assessed by means of force platforms. However, most of these devices are stationary, that is the patient is the dynamic element which can generate an evaluation with high subjectivity index. Therefore, this study aimed at developed a reaction force to the ground platform which provides mechanical stimuli controlled to quantify the distribution of the mass center as a function of the angular variation in the elderly ankle in the upright position. The construction of the prototype was divided into 3 steps, based on the two-dimensional movement of the ankle joint. In the 1st stage the construction of the mechanical assembly; in the 2nd stage development of the electronics; and 3rd stage the development of the supervisory system (control system). The force plataform was evaluated following the engineering functional tests such as: characterization and calibration of the sensors, the definition of the transfer function and accuracy of tests of angular movements (+ 10 ° and -10 ° to the movements of inversion and eversion, + 15 and -15º to the movements of dorsiflexion and plantar flexion). For the tests with volunteers were selected 30 volunteers.

ELIGIBILITY:
Inclusion Criteria:

* We included in this study individuals male and female
* Age ranging from 20 to 85 years
* Asymptomatic individuals
* Must walk without the use of an attachment
* Do not present motor deficit that makes the study impossible

Exclusion Criteria:

* Decompensated congestive heart failure
* Neurological or neurological diseases that interfere with significant neuromotor
* Individuals who did not agree to participate in the study

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 30 individuals, asymptomatic
Enrollment: 30 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-07-20 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Mass distribution | 15 minutes
  The center of mass was measured by the patient remaining on the force platform, remaining for 10 seconds in each angulation variant Unit of measurement: Kilograms (kg)

IPD SHARING:
Plan to Share IPD: No